CLINICAL TRIAL: NCT02878278
Title: Research About the Differences Between Chidamide Taken Daily and Twice a Week in Pharmacokinetics
Brief Title: Differences Between Chidamide Taken Daily and Twice a Week in Therapeutic Effect，Pharmacokinetics, Pharmacodynamics and EB Virus Activation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huiqiang Huang (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, Doctor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sunyat-senU201602101
Record Dates: First submitted 2016-08-20; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma, Extranodal NK-T-Cell; EBV
Keywords: Chidamide; Administration method
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chidamide BIW (Experimental): Chidamide is given 30mg,5mg/pill,twice a week, for at least 6 weeks
  Interventions: Drug: Chidamide BIW
- Chidamide QD (Experimental): Chidamide is given 10mg,5mg/pill, everyday,for at least 6 weeks.
  Interventions: Drug: Chidamide QD

INTERVENTIONS:
Drug: Chidamide BIW — Chidamide is given 30mg, twice a week
  Other Names: Epidaza
  Arms: Chidamide BIW
Drug: Chidamide QD — Chidamide is given 10mg,QD
  Other Names: Epidaza
  Arms: Chidamide QD

SUMMARY:
1. To compare the therapeutic effects, safety and the corresponding pharmacokinetics and pharmacodynamics between two different method of drug administration: 10mg, daily and 30mg/d, twice every week, and find out the more effect way of Chidamide administration.
2. To examine whether Chidamide could activate EB virus, and whether the above two different ways of administration are different in EB virus activation.

DETAILED DESCRIPTION:
Currently, Chidamide is taken twice a week, this comes from cell experiment and phase I clinical trial, which showed that the de-acetylation effect of Chidamide could last for 72 hours after administration. However, daily administration of Chidamide may create a more steady Chidamide concentration, thus improve the de-acetylation effect of Chidamide, so it's necessary to compare the two different ways of administration.

Current study showed that Romidepsin, a HDACI, could activate EBV during the treatment of NKTCL, whether Chidamide, as a novel HDACI, could activate EBV is still not clear, so this problem is worth to be accessed.

ELIGIBILITY:
Inclusion Criteria:

1. NKTCL patients confirmed by histopathology examination.
2. Age 18-75 years old, male or female, fertile women should have effective contraceptive measures.
3. NT/T cell lymphoma patients with disease progression or non-remission after L-asparaginase treatment or L-asparaginase-contained regimen treatment. Non-remission is defined as: patients do not have partial remission (PR) or better responses after treated by L-asparaginase contained regimen.
4. Patients who had 1-3 regimens (including chemotherapy, stem cell transplantation), but did not achieve remission or relapsed after remission.
5. With at least 1 measurable focus, whose long diameter ˃ 1.5cm, short diameter ˃1.0cm, or at least one evaluable focus.
6. Body weight: male 67±20 kilograms (47-87 kg), female 55±20 kilograms (35-75 kg);
7. Blood-routine test within 14 days of enrollment should satisfy (except lymphoma-related abnormalities): Hb≥80g/L，ANC≥1.0×109/L，PLT≥75×109/L；
8. ECOG: 0-2;
9. Estimated survival ≥ 3 months;
10. Willing to sign the written consent before the trial.

Exclusion Criteria:

1. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures.
2. QTc elongation with clinical significance ( male˃ 450ms, female˃ 470ms), ventricular tachycardia, atrial fibrillation, cardiac conducting blockage, myocardial infarction within 1 year, congestive heart failure, symptomatic coronary heart disease that requires treatment.
3. Cardiac B ultrasound show end-diastolic pericardial dark zone≥ 10cm
4. Patients who have received organ transplantation.
5. Patients received symptomatic treatment for bone marrow toxicity within 7 days prior to enrollment.
6. Patients with active hemorrhage.
7. Patients with or with history of thrombosis, embolism, cerebral hemorrhage, or cerebral infarction.
8. Patients with active infection, or with continuous fever within 14 days prior to enrollment.
9. Had major organ surgery within 6 weeks prior to enrollment.
10. Abnormal blood routine test results within 14 days prior to enrollment (Hb˂80g/L，ANC˂1.0×109/L，PLT˂75×109/L； Impaired liver function ( Total bilirubin ˃ 1.5 times of normal maximum, ALT/AST˃ 2.5 times of normal maximum, for patients with infiltrative liver disease ALT/AST ˃ 5 times of normal maximum), impaired renal function (serum creatinin˃ 1.5 times of normal maximum).
11. Patients with history of Chidamide treatment and had disease progression within 6 months afterward;
12. Patients that received large dose of steroids (˃10mg/d dexamethasone or other steroids of the equivalent dosage) within 4 weeks prior to enrollment;
13. Patients with hemophagocytic syndrome;
14. Patients with central nerve system diseases or history of central nerve system diseases;
15. Patients with mental disorders or those do not have the ability to consent;
16. Patients that had been enrolled in other clinical trials within 3 months prior to enrollment;
17. Patients with drug abuse, long term alcoholism that may impact the results of the trial.
18. Non-appropriate patients for the trial according to the judgment of the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | through study completion, an average of 30 months
Duration of Response (DOR) | through study completion, an average of 30 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | through study completion, an average of 30 months
Overall Survival (OS) | through study completion, an average of 30 months
EBV-DNA | through study completion, an average of 30 months
EBV-antibodies | through study completion, an average of 30 months
white blood cell count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
red blood cell count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood Hb level | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood platelet count | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
vital signs | every week though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum alanine aminotransferase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum aspartate transaminase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum total bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum direct bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum indirect bilirubin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum glutamyltranspeptidase level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum albumin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum ureal nitrogen level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
Serum creatinin level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
fasting blood glucose level | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood electrolytes level（K+, Na+，Cl-，Ca2+，Mg2+） | every 3 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
blood LDH level | every 6 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months
QTc from ECG | every 6 weeks though study completion，from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months

IPD SHARING:
Plan to Share IPD: Yes
The data of the trial would be accessable on the corresponding website after the trial is finished.

REFERENCES:
- [Derived] Chen J, Zuo Z, Gao Y, Yao X, Guan P, Wang Y, Li Z, Liu Z, Hong JH, Deng P, Chan JY, Cheah DMZ, Lim J, Chai KXY, Chia BKH, Pang JWL, Koh J, Huang D, He H, Sun Y, Liu L, Liu S, Huang Y, Wang X, You H, Saraf SA, Grigoropoulos NF, Li X, Bei J, Kang T, Lim ST, Teh BT, Huang H, Ong CK, Tan J. Aberrant JAK-STAT signaling-mediated chromatin remodeling impairs the sensitivity of NK/T-cell lymphoma to chidamide. Clin Epigenetics. 2023 Feb 6;15(1):19. doi: 10.1186/s13148-023-01436-6. PMID 36740715